CLINICAL TRIAL: NCT06379750
Title: STOP NCDs: Scaling Up Evidence-based Health System Interventions Through the Use of Sustainable Healthcare Financing and Digital TechnOlogy Platforms to Improve Non- Communicable Disease Prevention and Control in Tanzania
Brief Title: Using Healthcare Financing and Digital Technology to Improve Hypertension Prevention and Control in Tanzania
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Kilimanjaro Clinical Research Institute (Other); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Dr. Karen Yeates, Professor, Queen's University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: STOPNCD
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Diabetes
Keywords: hypertension; diabetes; NCD management; NCD prevention; mHealth; healthcare financing
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Enhanced Usual Care (EUC) (No Intervention): Enhanced usual care provided by facility MD or equivalent (control group)
- EUC + community support (Active Comparator): Enhanced usual care AND community-based peer-support model using WelTel check-ins and BCC SMS and facilitated group self monitoring
  Interventions: Other: Community-based peer-support model
- EUC + nurse-delivered check ins (Active Comparator): Enhanced usual care AND nurse-delivered HTN, DM and CVD risk assessment, diagnosis and Management using WelTel check-ins and BCC SMS
  Interventions: Other: Nurse-delivered care using WelTel check-ins and BCC SMS
- EUC + community support + nurse-delivered check ins (Active Comparator): Enhanced usual care AND nurse-delivered HTN, DM and CVD risk assessment, diagnosis and Management using WelTel check-ins and BCC SMS AND community-based peer-support model using WelTel check-ins and BCC SMS and facilitated group self monitoring
  Interventions: Other: Nurse-delivered care using WelTel check-ins and BCC SMS; Other: Community-based peer-support model

INTERVENTIONS:
Other: Nurse-delivered care using WelTel check-ins and BCC SMS — Nurse-delivered HTN, DM and CVD risk assessment, diagnosis and Management (through NIMONCD) using WelTel check-ins and BCC SMS
  Arms: EUC + community support + nurse-delivered check ins; EUC + nurse-delivered check ins
Other: Community-based peer-support model — Community-based peer- support model using Weltel check-ins and BCC SMS and facilitated group self monitoring
  Arms: EUC + community support; EUC + community support + nurse-delivered check ins

SUMMARY:
The aim of our proposed program is to develop and implement a multilevel, multicomponent and health-financing intervention that will facilitate the scale up of evidence-based strategies to improve non-communicable diseases prevention, detection and control in Tanzania. The investigators will accomplish this by: 1) adapting two intervention components that are candidates for inclusion in a highly effective optimized strategy (called STOP-NCDs) and; (b) Assess their individual and combined effectiveness and 2) conducting a robust, mixed-methods evaluation of the implementation process and assess factors that may influence implementation and sustainability for delivering and scaling the optimized STOP-NCDs strategy. The investigators will select and/or adapt intervention components making up the optimized STOP-NCDs strategy. Using a hybrid clinical-effectiveness implementation design, the investigators will conduct a study in 2 sequential phases: 1) A clinical-effectiveness phase in which the investigators evaluate the effect of our combined strategies (task-sharing and WelTel) versus Usual Care, on rates of systolic BP reduction at 12 months; as well as other secondary outcomes including diagnosis and treatment of diabetes and, patient knowledge of CVD risks and prevention, and, other features of health provider NCD prevention activities. 2) A post-implementation phase in which the investigators use the RE-AIM framework to evaluate changes in the adoption and maintenance of our combined strategies in participating iCHF health facilities across Kilimanjaro region. The investigators will use the WelTel communication and Patient Management platform for to deliver culturally and contextually appropriate evidence-based text messaging to patients. It allows for quality improvement and is a unique tool for our program to scaling low-cost interventions that provide capabilities for tracking of health system service uptake, quality-metrics at health facilities, drug stock-out management, and patient-centered behavioral health interventions. Deployment of WelTel will allow for integration of NCD prevention targeted health services to all adult iCHF members across differing life stages and NCD risk and have a significant impact on increasing quality of care and sustainability of health financing and performance-based incentives through improved prescribing, patient engagement, medication adherence and healthy behaviour change.

ELIGIBILITY:
Inclusion Criteria:

* All adults with uncontrolled HTN who receive care through iCHF membership and are able to provide informed consent.

Exclusion Criteria:

* Adults with controlled HTN or those without a diagnosis of HTN
* Unable or unwilling to provide informed consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1320 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 12 months
  Change in systolic blood pressure from baseline to last follow-up visit

SECONDARY OUTCOMES:
Blood pressure control | 12 months
  Proportion of participants with controlled blood pressure (<140 mm Hg for systolic and <90 mm Hg for diastolic) at the last follow-up visit